CLINICAL TRIAL: NCT05605483
Title: Salad Bars in the National School Lunch Program: Impact on Dietary Consumption Patterns in Elementary School Students
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: George Mason University (Other); University of North Carolina, Chapel Hill (Other); The University of Tennessee, Knoxville (Other)
Responsible Party: Sponsor
Other Study IDs: HM20012226
Record Dates: First submitted 2022-10-28; First posted 2022-11-04 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Diet, Food, and Nutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Schools with salad bars: Schools with salad bars
  Interventions: Other: Salad bar
- Schools without salad bars: Schools without salad bars
  Interventions: Other: Waitlisted control
- Schools with salad parts post COVID-19: A subset schools with salad bars that were examined pre-COVID-19 will undergo methods again.
  Interventions: Other: Salad bar post-COVID

INTERVENTIONS:
Other: Salad bar — Schools where the school district has installed salad bars
  Groups: Schools with salad bars
Other: Waitlisted control — Schools where the school district has not yet installed salad bars
  Groups: Schools without salad bars
Other: Salad bar post-COVID — Schools where the school distract has re-opened salad bars will have methods repeated in a subset of schools post-COVID-19
  Groups: Schools with salad parts post COVID-19

SUMMARY:
This project is a research study looking at what foods students choose and eat during school lunch and examines how salad bars impact what children eat.

DETAILED DESCRIPTION:
This project applies a wait list control cluster randomized controlled trial to evaluate school salad bars. This project uses digital images (pictures) of labeled trays in the cafeteria before and after children eat lunch. This project also asks cafeteria workers about their thoughts about salad bars and their experiences with the salad bar program.

ELIGIBILITY:
Inclusion Criteria:

* Students: All K-6th grade students at target schools who participate in the school lunch program on rating day
* Cafeteria staff: All cafeteria personnel at the randomly selected target schools will be eligible to complete surveys

Exclusion Criteria:

* Students: Unsure sex of child
* Cafeteria staff: None

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All K-6th students who participate in the school lunch program and all cafeteria personnel at target schools
Sampling Method: Non-Probability Sample
Enrollment: 6269 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
fruits and vegetables (FV) selection | Baseline to up to 6 weeks after salad bars installed
  Amount of FV selection will be calculated based on digital photographs of student's lunch trays before consumption
FV consumption | Baseline to up to 6 weeks after salad bars installed
  Amount of FV consumed will be calculated by subtracting amount of FV remaining after lunch is consumed from amount of FV selected based on digital photographs of student's lunch trays before and after consumption.

SECONDARY OUTCOMES:
energy intake (kcal) | Baseline to up to 6 weeks after salad bars installed
  Amount of calories consumed will be calculated by subtracting the total amount of calories remaining on trays from the total amount of calories initially selected based on digital photographs of student's lunch trays before and after consumption.
dietary quality (Healthy Eating Index) | Baseline to up to 6 weeks after salad bars installed
  the Healthy Eating Index will be calculated for food and beverages consumed at lunch (amount on the tray before minus after consumption) using NDSR
fruits and vegetables (FV) selection post-COVID-19 | 4-6 weeks after salad bars re-installed
  To examine the the impact of salad bars on student dietary intake patterns after their reintroduction post-COVID-19 school closures. Amount of FV selection will be calculated based on digital photographs of student's lunch trays before consumption
FV consumption post-COVID-19 | 4-6 weeks after salad bars re-installed
  To examine the the impact of salad bars on student dietary intake patterns after their reintroduction post-COVID-19 school closures. Amount of FV consumed will be calculated by subtracting amount of FV remaining after lunch is consumed from amount of FV selected based on digital photographs of student's lunch trays before and after consumption.
energy intake (kcal) post-COVID-19 | 4-6 weeks after salad bars re-installed
  To examine the the impact of salad bars on student dietary intake patterns after their reintroduction post-COVID-19 school closures. Amount of calories consumed will be calculated by subtracting the total amount of calories remaining on trays from the total amount of calories initially selected based on digital photographs of student's lunch trays before and after consumption.
dietary quality (Healthy Eating Index) post-COVID-19 | 4-6 weeks after salad bars re-installed
  To examine the the impact of salad bars on student dietary intake patterns after their reintroduction post-COVID-19 school closures. The Healthy Eating Index will be calculated for food and beverages consumed at lunch (amount on the tray before minus after consumption) using NDSR

CONTACTS AND LOCATIONS:
Overall Officials: Melanie K Bean, PhD, Principal Investigator — VCU
Locations (1):
- Healthy Lifestyles Center at the Children's Hospital of Richmond at VCU, Henrico, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bean MK, Mazzeo SE, de Jonge L, Thornton L, Raynor H, Mendoza A, Farthing S, Moore B. Impact of school salad bars on fruit and vegetable selection, intake, and waste in Mid-Atlantic elementary schools. Int J Behav Nutr Phys Act. 2025 Feb 5;22(1):15. doi: 10.1186/s12966-025-01713-y. PMID 39910590
- [Derived] Bean MK, Raynor HA, Thornton LM, de Jonge L, Mazzeo SE. Design and rationale for evaluating the impact of salad bars on elementary school students' fruit, vegetable, and energy intake: a wait list control, cluster randomized controlled trial. BMC Public Health. 2022 Dec 9;22(1):2304. doi: 10.1186/s12889-022-14744-y. PMID 36494649